CLINICAL TRIAL: NCT05159154
Title: Myocardial Work in Septic Shock Patients: an Observational Study
Brief Title: Myocardial Work in Septic Shock Patients
Acronym: MYWORKSS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Humanitas Clinical and Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: MYWORKSS
Record Dates: First submitted 2021-12-03; First posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Septic Shock; Critical Illness
MeSH Terms: conditions — Shock, Septic; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Septic Shock Patients: Patients admitted with diagnosis of septic shock
  Interventions: Device: Myocardial Work

INTERVENTIONS:
Device: Myocardial Work — Myocardial work (MW) is emerging as an alternative tool for studying LV myocardial systolic function, because it incorporates both deformation and load into its analysis. In this context, MW could be considered as an advancement of myocardial strain, allowing to investigate LV performance also in cases of changes in afterload that could lead to misleading conclusions if relying only on strain analysis. This parameter will be evaluated by using an echographer equipped with a specific software for the analysis (Ecog Vivid E95 Ultra GE®)

SUMMARY:
Myocardial strain analysis has emerged in the last decade as a reliable tool for studying myocardial mechanics, adding information on cardiac performance when compared with traditional parameters of left ventricle (LV) systolic function, such as ejection fraction (EF).

However, their relative load dependency makes the myocardial deformation indices unable to account for changes in pre- and afterload.

Myocardial work (MW) is emerging as an alternative tool for studying LV myocardial systolic function, because it incorporates both deformation and load into its analysis.

The purpose of this observational trial is to validate the use of MW in septic shock patients by means of consecutive echocardiographic assessment at predefined timepoints. Secondarily, we'll evaluate the impact of the vasoactive drugs used in septic shock patients (vasopressors and inotropes) on MW and on ventriculo-arterial coupling.

DETAILED DESCRIPTION:
Myocardial strain analysis has emerged in the last decade as a reliable tool for studying myocardial mechanics, adding information on cardiac performance when compared with traditional parameters of left ventricle (LV) systolic function, such as ejection fraction (EF).

However, their relative load dependency makes the myocardial deformation indices unable to account for changes in pre- and afterload.

Myocardial work (MW) is emerging as an alternative tool for studying LV myocardial systolic function, because it incorporates both deformation and load into its analysis. In this context, MW could be considered as an advancement of myocardial strain, allowing to investigate LV performance also in cases of changes in afterload that could lead to misleading conclusions if relying only on strain analysis.

Conditions of increased afterload can in fact negatively impact on myocardial strain even if MWis normal. MW assessment was initially calculated using invasive pressure measurements, which limited its widespread use in clinical practice.

Recently, Russell et al. demonstrated that pressure-strain loops (PSLs) could estimate LV performance in a non-invasive manner, deriving LV pressure (LVP) curves from non-invasively acquired brachial artery cuff pressure. To date, the technique has been applied in myocardial ischaemia and in identification of cardiac resynchronization therapy (CRT)-responders with good results.

This clinical approach has been never tested, insofar, septic shock patients. The heart is one of the organs most frequently failing in sepsis; however, depending on the definition used, the prevalence of sepsis-induced cardiac dysfunction may vary between 10% and 70%. The sepsis-induced dysregulated inflammatory response has been directly linked to cardiomyocyte dysfunction, leading to a broad spectrum of cardiomyopathies, including ventricles' impairment during systole or diastole, inadequate cardiac output, oxygen delivery, or primary myocardial cellular injury.

Hence, in septic shocked patients, echocardiography plays a pivotal role, identifying most of the clinical cardiac patterns related to acute systolic dysfunction and chambers' dilation using basic level 2D and M-mode echocardiography. A more comprehensive diagnosis can be achieved with advanced levels of competency. Simultaneously, hemodynamic evaluation and monitoring are possible with advanced levels of competency, including the use of color Doppler, spectral Doppler, tissue Doppler imaging, and, eventually, 3D or speckled tracking. Specific pathways can now achieve all these steps of competence for skills certification, developed by intensive care medicine societies.

A variety of cardiac changes can be associated with septic shock, although a normal study is not unusual [7]. Abnormalities in LVEF (i.e., contractile impairment may be associated with either a global dysfunction or exhibited as specific patterns with apical akinesis and ballooning accompanied by good basal LV contraction and is almost always reversible over days), LV diastolic function, and right ventricular (RV) function have all been described. Since the resuscitation in septic shock is mainly focused on an aggressive and rapid fluid resuscitation associated with the administration of systemic vasopressors to optimize cardiac preload, output, and peripheral perfusion, the assessment of the basal cardiac function is critical and should be routinely performed at the bedside for this purpose.

The dynamic interaction between the heart and the systemic circulation allows the cardiovascular system to be efficient in providing adequate cardiac output and arterial pressures necessary for sufficient organ perfusion. The cardiovascular system provides adequate pressure and flow to the peripheral organs in different physiological and pathological conditions because of the continuous modulation of the arterial system compliance, stiffness and resistance with respect to LV systolic performance. This challenging interplay may lead to a condition called "ventriculo-arterial uncoupling", when the ration between myocardial performance and peripheral response (Ea/Ees) is unbalanced. The hemodynamic profile of septic shock is primarily characterized by generalized vasodilatation resulting in severe hypotension with systemic hypoperfusion. In most of the patients with septic shock, cardiovascular efficiency is impaired, and the Ea/Ees becomes uncoupled (Ea/Ees > 1). Th e hemodynamic profile is characterized by both the significant increase in Ea and the decrease in Ees. Because the increase in Ea is generally induced by pharmacological vasoconstriction. (norepinephrine) and the consequent increase in arterial tone, a decrease in Ees generally depends on the reduction in myocardial contractility. Whatever the underlying mechanism, when A-V uncoupling occurs in septic shock, the cardiac energetics are unfavorable and are often sacrificed to maintain tissue perfusion.

The purpose of this observational trial is to validate the use of MW in septic shock patients by means of consecutive echocardiographic assessment at predefined timepoints. Secondarily, we'll evaluate the impact of the vasoactive drugs used in septic shock patients (vasopressors and inotropes) on MW and on ventriculo-arterial coupling.

ELIGIBILITY:
Inclusion criteria:

* Expected to be ventilated for > 48 hours
* Age > 50

Exclusion criteria:

* Atrial fibrillation (at the admission or during intensive care unit stay);
* Neuromuscular disorders;
* Home ventilation prior to admission;
* Palliative intubation;
* Intubation for an indication to tracheostomy;
* Poor acoustic window (after the first assessment);
* Severe mitral and/or aortic valve stenosis or regurgitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of septic shock < 24h and acute circulatory failure was defined as at least one of the following criteria:
  * Systolic arterial pressure ≤ 90 mmHg (or a decrease > 50 mm Hg in hypertensive patients) or a mean arterial pressure (MAP) ≤ 70 mmHg or the use of vasopressors to maintain SAP > 90 mmHg.
  * skin mottling
  * tachycardia ≥100 beats/min
  * urinary flow ≤ 0.5 mL/kg for at least 2 hours
  * blood lactate level ≥ 2 mmol/L.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Myocardial Work | 24h from intensive care unit admission
  Quantification of Myocardial Work Index

SECONDARY OUTCOMES:
Myocardial Work | 60 +/- 12 h from intensive care unit admission
  Quantification of Myocardial Work Index
Myocardial Work | 7 days from intensive care unit admission
  Quantification of Myocardial Work Index

OTHER OUTCOMES:
Myocardial Work | 1h from norephinefrine infusion start
  Quantification of Myocardial Work Index
Myocardial Work | 1h from norephinefrine infusion dose increase
  Quantification of Myocardial Work Index
Myocardial Work | 6h from norephinefrine infusion dose increase
  Quantification of Myocardial Work Index
Myocardial Work | 1h from dobutamine infusion start
  Quantification of Myocardial Work Index

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Clinical and Research center, Rozzano, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided
The datasets used and/or analyzed during the current study are available from the corresponding author on reasonable request